CLINICAL TRIAL: NCT07385313
Title: Randomized Prospective Evaluation of Ovine Forestomach Matrix (OFM) and NPWT to Accelerate Tissue Coverage Over Exposed Structures
Brief Title: Combined OFM and Vacuum-assisted Therapy for Expedited Regeneration Over Structures
Acronym: COVER
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aroa Biosurgery Limited (Industry)
Collaborators: Coalition for National Trauma Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP.AROA.005
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Defects; Soft Tissue Wounds; Traumatic Soft Tissue Defect
Keywords: Traumatic Wounds; Soft Tissue Repair; Negative Pressure Wound Therapy; Ovine Forestomach Matrix; Wound Healing
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two arms:
  * Interventional Arm: Myriad™ applied in conjunction with NPWT ('Myriad+NPWT')
  * Control Arm: NPWT alone ('NPWT')
Masking Description: Investigators cannot be blinded to the treatment groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Interventional Arm (Experimental): Myriad™ applied in conjunction with NPWT ('Myriad+NPWT')
  Interventions: Device: Myriad™ applied in conjunction with NPWT
- Control Arm (Active Comparator): NPWT alone ('NPWT')
  Interventions: Device: NPWT Alone

INTERVENTIONS:
Device: Myriad™ applied in conjunction with NPWT — Myriad™ applied in conjunction with NPWT ('Myriad+NPWT')
  Arms: Interventional Arm
Device: NPWT Alone — Control Arm: NPWT alone ('NPWT')
  Arms: Control Arm

SUMMARY:
Demonstrate faster tissue coverage of exposed structures using OFM in combination with negative pressure wound therapy (NPWT), versus NPWT alone

DETAILED DESCRIPTION:
Ovine forestomach matrix (OFM) is a decellularized extracellular matrix bioscaffold developed for a range of soft tissue repair, reconstruction, and wound healing applications. OFM is a platform technology used in numerous products, including Myriad™ Matrix, Endoform™ Natural, Endoform™ Antimicrobial, and Ovitex® Reinforced Bioscaffolds. Preclinical and clinical studies have evaluated OFM with respect to mesenchymal stromal cell recruitment, cellular proliferation, angiogenesis, vascularization, and modulation of wound protease activity. Over time, the OFM material is resorbed and incorporated into the patient's soft tissue during the wound healing process.

Myriad devices are composed entirely of OFM and are available in either a sheet ("Matrix") or particulate ("Morcells") configuration. The devices are applied directly to soft tissue defects to support tissue infill and coverage. These devices have been the subject of multiple clinical studies across a spectrum of applications in wound healing, soft tissue repair, and plastic and reconstructive surgery. These studies, together with extensive preclinical testing, provide background information regarding the use of Myriad devices across a range of procedures in the general patient population.

The present study has been designed as a randomized clinical investigation to evaluate outcomes associated with the use of Myriad devices in the treatment of traumatic wounds when used in combination with negative pressure wound therapy (NPWT). Myriad devices are indicated for soft tissue repair and reconstruction and may be used at the discretion of the attending physician. Myriad devices may be used concomitantly with NPWT across a wide range of surgical procedures where soft tissue is missing or damaged.

This randomized clinical investigation design has been selected to generate additional clinical evidence to evaluate time (in days) to achieve complete tissue coverage of exposed structures, wound volume reduction, wound area reduction, and other key clinical parameters in traumatic wound management.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered eligible for the study based on the following criteria:

  * Willing and able to provide written informed consent and to comply with the requirements of the Clinical Investigational Plan
  * Male or female patients aged 18 years or above
  * Patient is requiring reconstruction of a full thickness soft tissue defect, that includes exposed structures (bone, tendon, or neurovascular), upper or lower extremity.
  * Total defect size, range 25 to 800 cm2

Exclusion Criteria:

* Patients will be excluded from the study based on the following criteria:

  * Patients with known sensitivity to ovine (sheep) derived material
  * Pregnant or lactating females.
  * Patients who are prisoners.
  * Patients who are likely not to complete the study.
  * Patients who, in the opinion of the Investigator, are unlikely to comply with the protocol.
  * Patients currently participating in or have participated in another clinical study within the past 30 days prior to enrolment that at the discretion of the Investigator makes them unsuitable for inclusion in the study.
  * Any subject who, at the discretion of the Investigator, is not suitable for inclusion in the study.
  * Any medical condition, recent treatment or serious intercurrent illness that, in the opinion of the Investigator, may make it undesirable for the patient to participate in the study.
  * Obesity (BMI>45)
  * Blood glucose ≥350 mg/dL at admission
  * History of chronic peripheral vascular disease
  * Current immunosuppression
  * Recent neoadjuvant chemotherapy or radiotherapy
  * Previous or concurrent application of a cell/tissue-based product (CTP, or skin substitute) at the wound site within 30 days of the Screening Visit
  * Defect is a third degree burn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Tissue Coverage | Up to 56 days/ 8 week follow up
  Time (days) to complete tissue coverage of the exposed structure

SECONDARY OUTCOMES:
Complete coverage of exposed structures | up to 28 days (4 weeks)
  Percent of defects with complete coverage of exposed structures by 4 weeks
Post operative complications | Up to 56 days/ 8 week follow up
  Percent of patients with post operative complications (defined as seroma, hematoma, minor infection (cellulitis), major infection (requiring additional surgical intervention, incision and drainage, debridement, additional usage of/change in antibiotic therapy), or skin necrosis/dehiscence)
NPWT Usage | Up to 56 days/ 8 week follow up
  Length of Negative Pressure Wound Therapy (NPWT) usage (days)
Wound depth infill | 56 days/up to 8 weeks
  Rate of depth infill (mm per week)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Rizzo, MD, Principal Investigator — Brooke Army Medical Center
Locations (2):
- United States (2):
  - University of Colorado-Anschutz Medical Campus, Aurora, Colorado
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available one year after initial results publication.